CLINICAL TRIAL: NCT03705169
Title: A Phase I, First-in-Human Study of SAR441236, a Tri-specific Broadly Neutralizing Antibody, in Participants With HIV
Brief Title: Pharmacokinetics and Safety of SAR441236
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study closed to enrollment and follow-up in May 2023. There had been no enrollment since October 2021, and by 2023, the available study product had reached its expiration date. Enrollment targets in Arm B had not been met.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sanofi (Industry); ModeX Therapeutics, An OPKO Health Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5377; 38508 (Registry Identifier: DAIDS-ES Registry Number); TDU15867 (Other: Sanofi)
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: HIV-1-infection
Keywords: HIV; pharmacokinetics; pharmacodynamics; broadly neutralizing antibody; antiretroviral; Phase 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Arm A: 1 mg/kg SAR441236 (Experimental): Participants continued on non-study-provided ART and received 1 mg/kg of SAR441236, administered as a single intravenous (IV) infusion on Day 0 (Cohort 1).
  Interventions: Biological: SAR441236
- Arm A: 3 mg/kg for SAR441236 (Experimental): Experimental: Arm A: 3 mg/kg SAR441236 Participants continued on non-study-provided ART, and received 3 mg/kg of SAR441236, administered as a single IV infusion on Day 0 (Cohort 2).
  Interventions: Biological: SAR441236
- Arm A: 10 mg/kg SAR441236 (Experimental): Participants continued non-study-provided ART and received 10 mg/kg of SAR441236, administered as a single IV infusion on Day 0 (Cohort 3).
  Interventions: Biological: SAR441236
- Arm A: 30 mg/kg SAR441236 (Experimental): Participants continued non-study-provided ART and received 30 mg/kg of SAR441236, administered as an IV infusion on Day 0 and then every 12 weeks for a total of four doses (Cohort 4).
  Interventions: Biological: SAR441236
- Arm A: 0 mg/kg SAR441236 (Placebo Comparator): Placebo participants were pooled across those receiving:
  * 1 mg/kg dose volume-equivalent administered as a single IV infusion (Cohort 1).
  * 3 mg/kg dose volume-equivalent administered as a single IV infusion (Cohort 2).
  * 10 mg/kg dose volume-equivalent administered as a single IV infusion (Cohort 3)
  * 30 mg/kg dose volume-equivalent administered as an IV infusion on Day 0 and then every 12 weeks for a total of four doses (Cohort 4)
  All continued on non-study provided ART.
  Interventions: Biological: Placebo
- Arm B: 1 mg/kg SAR441236 (Experimental): Participants received 1 mg/kg of SAR441236, administered as a single IV infusion on Day 0. Antiretroviral treatment was initiated or re-initiated by Day 28 (Cohort 5).
  Interventions: Biological: SAR441236
- Arm B: 30 mg/kg SAR441236 (Experimental): Participants received 30 mg/kg of SAR441236, administered as a single IV infusion on Day 0. Antiretroviral treatment was initiated or re-initiated by Day 28 (Cohort 8).
  Interventions: Biological: SAR441236
- Arm C: 0.3 mg/kg SAR441236 (Experimental): Participants continued non-study-provided ART and received 0.3 mg/kg of SAR441236, administered as a subcutaneous (SC) injection(s) on Day 0 (Cohort 10).
  Interventions: Biological: SAR441236
- Arm C: 1 mg/kg SAR441236 (Experimental): Participants continued non-study-provided ART and received 1 mg/kg of SAR441236, administered as an SC injection(s) on Day 0 (Cohort 11).
  Interventions: Biological: SAR441236
- Arm C: 0 mg/kg SAR441236 (Placebo Comparator): Placebo participants were pooled across those receiving:
  * 0.3 mg/kg dose volume-equivalent administered as an SC injection(s) (Cohort 10).
  * 1 mg/kg dose volume-equivalent administered as an SC injection(s) (Cohort 11).
  All continued on non-study provided ART.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SAR441236 — Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
  Arms: Arm A: 1 mg/kg SAR441236; Arm A: 10 mg/kg SAR441236; Arm A: 3 mg/kg for SAR441236; Arm A: 30 mg/kg SAR441236; Arm B: 1 mg/kg SAR441236; Arm B: 30 mg/kg SAR441236; Arm C: 0.3 mg/kg SAR441236; Arm C: 1 mg/kg SAR441236
Biological: Placebo — Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
  Arms: Arm A: 0 mg/kg SAR441236; Arm C: 0 mg/kg SAR441236

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of SAR441236, a tri-specific broadly neutralizing antibody against the human immunodeficiency virus (HIV).

DETAILED DESCRIPTION:
This study evaluated the safety, tolerability, pharmacokinetics, and antiviral activity of SAR441236, a tri-specific broadly neutralizing antibody against HIV.

The study included three arms.

In Arm A, three dose cohorts (1, 3, and 10 mg/kg) of antiretroviral-treated, virologically suppressed participants were randomized (2:1, active to placebo) to receive a single intravenous (IV) dose of SAR441236 or placebo on Day 0. After Cohort 1 (1 mg/kg, lowest Arm A dose), each subsequent, higher-dose, cohort opened for enrollment only after an evaluation of safety outcomes for all participants in the previous cohort indicated it was safe to increase the dose of SAR441236. All participants in Cohorts 1-3 were followed for up to 24 weeks.

In Arm A, Cohort 4, participants were randomized (2:1, active to placebo) to receive an IV infusion of 30 mg/kg SAR441236 or placebo once every 12 weeks beginning at entry, for a total of 4 infusions. The first six Cohort 4 participants were enrolled after the safety evaluation of Cohort 3 participants and the rest of the Cohort 4 participants were accrued after a safety evaluation of the first 6 participants. The time between infusions was prolonged for some participants due to the COVID-19 pandemic, which occurred during the course of the study. Participants in this cohort were followed for up to 36 weeks after their final infusion.

Participants in Arm A continued taking non-study-provided antiretroviral treatment throughout the study.

In Arm B, two cohorts of viremic participants received a single IV dose of SAR441236 on Day 0. Cohort 5 (1 mg/kg, lowest planned Arm B dose) opened first. After reviewing the safety data from that cohort, as well as that from all Arm A cohorts (which had fully enrolled), and taking into consideration enrollment challenges, the study was redesigned to be a dose de-escalation study in Arm B only. With this redesign, the study began enrollment into the highest dose (Cohort 8, 30 mg/kg) after closing Cohort 5 enrollment. Each subsequent Arm B cohort (of lower doses) was planned to open for enrollment only after an evaluation of efficacy data from Day 14 for all participants in the previous cohort was completed. However, the highest dose cohort never fully enrolled, and no subsequent cohorts were opened. All Arm B participants were followed for up to 24 weeks.

Participants in Arm B initiated or re-initiated non-study-provided combination antiretroviral therapy (ART) (selected by their primary HIV clinician) on or before Day 28. A later version of the protocol changed the duration of SAR441236 monotherapy to no more than 14 days, however, no participants enrolled under that version.

In Arm C, two cohorts of ART-treated, virologically suppressed participants were randomized (2:1, active to placebo) to receive a single subcutaneous (SC) dose of SAR441236 or placebo on Day 0. Cohort 11 (1 mg/kg) opened for enrollment only after an evaluation of safety outcomes from Day 14 for all participants in Cohort 10 (0.3 mg/kg) and the cumulative data from that cohort indicated it was safe to dose escalate. All Arm C participants were followed for 24 weeks.

Participants in Arm C continued taking non-study-provided ART throughout the study.

The study closed to enrollment and follow-up in May 2023 due to the expiration of the available study product, despite failing to meet its enrollment targets in Arm B. There had been no enrollment to the study since October 2021, despite the team's revision of the protocol (Version 4.0) to adjust eligibility criteria to facilitate enrollment of participants with viremia. At the time of study closure, Arm A and C were fully enrolled. Two Arm B cohorts (1 mg/kg and 30 mg/kg) achieved partial enrollment. Although protocol version 4.0 was released in September 2022, the last participant was enrolled under protocol version 3.0 and completed study follow-up in April 2022.

ELIGIBILITY:
Note: The following inclusion and exclusion criteria reflect those in protocol version 3.0, the last protocol version under which participants enrolled. Although a protocol version 4.0 was released, no participants enrolled under that version.

Inclusion Criteria, Arms A, B, and C

* HIV-1 infection, documented by any licensed rapid HIV-1 test or HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot, Geenius assay, or a second antibody test by a method other than the initial rapid HIV-1 and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

  * NOTE: The term "licensed" refers to a US Food and Drug Administration (FDA)-approved kit.
  * WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot, Geenius assay, or a plasma HIV-1 RNA viral load.
* The following laboratory values obtained within 45 days prior to entry by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.

  * Absolute neutrophil count (ANC) greater than or equal to 1500 cells/mm^3
  * Hemoglobin greater than or equal to 12.0 g/dL for men and greater than or equal to 11.0 g/dL for women
  * Platelet count greater than or equal to 120,000/mm^3
  * Creatinine clearance (CrCl) greater than 60 mL/min

    * Refer to the calculator located on the FSTRF website (at https://www.frontierscience.org/): Calculated Creatinine Clearance - Cockcroft-Gault Equation (Adult).
  * Aspartate aminotransferase (AST) (SGOT) less than 1.25 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) (SGPT) less than 1.25 x ULN
  * Alkaline phosphatase less than 2.0 x ULN
  * Total bilirubin less than 1.1 x ULN
* Hepatitis C virus (HCV) antibody negative result within 45 days prior to study entry or, for study candidates who are HCV antibody positive (based on testing performed at any time prior to study entry), a negative HCV RNA result obtained within 45 days prior to study entry.

  * NOTE: A negative HCV RNA level may result from either spontaneous clearance or from HCV therapy. Participants must have completed any HCV therapy at least 6 months prior to enrollment.
* Negative HBsAg result obtained within 45 days prior to study entry, or documented hepatitis B immunity, defined as positive hepatitis B surface antibody testing, at any time.
* Female study candidates of reproductive potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL performed at screening and again within 24 hours before study entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC)/CLIA-waived test.

  * NOTE: Reproductive potential is defined as girls who have reached menarche, and women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, and women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy.
* All study candidates must agree not to participate in an assisted conception process (e.g., sperm donation, intrauterine insemination, in vitro fertilization) from screening until 12 weeks after the final study visit.
* If participating in sexual activity that could lead to pregnancy, all study candidates must agree to use at least one reliable method of contraception from study entry until 12 weeks after the final study visit. At least one of the following methods must be used appropriately:

  * Condoms (male or female) with or without a spermicidal agent. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission.
  * Diaphragm or cervical cap with spermicide.
  * Intrauterine device.
  * Hormone-based contraceptive.
* Study candidates who are not of reproductive potential are eligible without requiring the use of a contraceptive method. Acceptable documentation of sterilization, menopause, and reproductive potential is specified below.

  * Written documentation or oral communication from a clinician or clinician's staff documented in source documents of one of the following:

    * Physician report/letter
    * Operative report or other source documentation in the patient record
    * Discharge summary
    * Laboratory report of azoospermia (is required to document successful vasectomy)
    * Follicle-stimulating hormone (FSH) measurement elevated into the menopausal range as established by the reporting laboratory.
  * NOTE A: Female reproductive potential is defined in the criteria above.
  * NOTE B: Male candidates who are not of reproductive potential are defined as having documented azoospermia.
  * NOTE C: A female study candidate's oral report of her male partner's lack of reproductive potential should be recorded in the source documents if written proof is not available.
* Ability and willingness of participant to provide informed consent.

Additional Arms A- and C-specific Inclusion Criteria

* Receiving combination ART for at least 12 months prior to study entry with no changes in ART regimen within the 12 weeks prior to entry.

  * NOTE A: Use of a two-drug ART regimen within the 12 months prior to entry is exclusionary.
  * NOTE B: Although ritonavir or cobicistat may be included in a combination ART regimen, neither of these "counts" in a tally of antiretroviral agents.
* CD4+ cell count of greater than or equal to 200 cells/mm^3 obtained within 45 days prior to study entry at any US laboratory that has a CLIA certification or its equivalent.
* Within 45 days prior to study entry, plasma HIV-1 RNA <50 copies/mL on any FDA-approved assay with a limit of quantification of <50 copies/mL by a US laboratory that has a CLIA certification or its equivalent.
* Within 12 months prior to study entry and before screening, at least one documented plasma HIV-1 RNA <50 copies/mL on any FDA-approved assay with a limit of quantification of <50 copies/mL by a US laboratory that has a CLIA certification or its equivalent.

  * NOTE: A single plasma HIV-1 RNA ≥50 but <200 copies/mL at least 6 months prior to screening is permitted if followed within 2 months by an HIV-1 RNA <50 copies/mL.

Additional Arm B-specific Inclusion Criteria

* Plasma HIV-1 RNA >5000 and ≤200,000 copies/mL within 45 days prior to study entry.
* CD4+ cell count of greater than or equal to 350 cells/mm^3 obtained within 45 days prior to study entry at any US laboratory that has a CLIA certification or its equivalent.
* Willingness and ability to start or re-start combination ART by or on Day 28 of the study.

Exclusion Criteria, Arms A, B, and C

* Breastfeeding or plans to become pregnant.
* Receipt of chimeric, humanized or human long-acting mAbs, whether licensed or investigational, within 12 months prior to entry, or receipt of chimeric, humanized or human regular mAbs, whether licensed or investigational, within 6 months prior to entry, unless reviewed and approved by the study's core team.
* Known allergy/sensitivity or any hypersensitivity to components of study treatment or its formulation (refer to the product's Investigator's Brochure).
* Vaccination within 30 days prior to entry or intent to receive an elective vaccination (e.g., hepatitis A vaccine, travel-related) during the course of the study except as noted in the study protocol.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 45 days prior to entry.
* Diagnosis of AIDS-defining illness using the current list on the US Centers for Disease Control and Prevention (CDC) website within 1 year prior to entry.
* Weight greater than 115 kg within 45 days prior to study entry.
* Use of maraviroc, ibalizumab, or enfuvirtide at any time.

Additional Arms A- and C-specific Exclusion Criterion

* Within 6 months prior to study entry, any plasma HIV-1 RNA ≥50 copies/mL on any FDA-approved assay with a limit of quantification of <50 copies/mL performed by a US laboratory that has a CLIA certification or its equivalent.

Additional Arm B-specific Exclusion Criterion

* Use of any anti-HIV ART, including FDA-approved pre-exposure prophylaxis (PrEP) within the preceding 3 months

Additional Arm C-specific Exclusion Criterion

* Presence of abdominal scarring or tattooing that could interfere with assessment of injection-site reaction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athe Tsibris, MD, MS, Study Chair — Brigham and Women's Hospital, Harvard Medical School; Daniel R. Kuritzkes, MD, Study Chair — Brigham and Women's Hospital Therapeutics CRS, Harvard Medical School; Pablo Tebas, MD, Study Chair — Penn Therapeutics CRS
Locations (23):
- United States (23):
  - Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - University of Washington Positive Research CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017. — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expediated Reporting of Adverse Events to DAIDS, Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 23 Clinical Research Sites (CRSs) in the United States between May 2019 and October 2021.
Pre-assignment Details: Participants who enrolled in Arms A and C were randomized 2:1 SAR441236:placebo. Participants who enrolled in Arm B were not randomized and were assigned open-label SAR4412326. For analysis, participants receiving placebo (of any dose-volume equivalent) are pooled within arm per the pre-specified analysis plan.
Groups:
- Arm A: 0 mg/kg SAR441236: Placebo participants were pooled across those receiving:
  * 1 mg/kg dose volume-equivalent administered as a single IV infusion (Cohort 1).
  * 3 mg/kg dose volume-equivalent administered as a single IV infusion (Cohort 2).
  * 10 mg/kg dose volume-equivalent administered as a single IV infusion (Cohort 3)
  * 30 mg/kg dose volume-equivalent administered as an IV infusion on Day 0 and then every 12 weeks for a total of four doses (Cohort 4)
  All continued on non-study provided ART.
  Placebo: Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
- Arm C: 0 mg/kg SAR441236: Placebo participants were pooled across those receiving:
  * 0.3 mg/kg dose volume-equivalent administered as an SC injection(s) (Cohort 10).
  * 1 mg/kg dose volume-equivalent administered as an SC injection(s) (Cohort 11).
  All continued on non-study provided ART.
  Placebo: Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
Period: Overall Study
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm A: 0 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236 | Arm C: 0 mg/kg SAR441236
Started | 4 | 4 | 4 | 11 | 10 | 5 | 2 | 4 | 4 | 4
Participants Receiving First Dose | 4 | 4 | 4 | 10 | 10 | 5 | 2 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 5 | 10 | 3 | 1 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 6 | 0 | 2 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Closure | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive study treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Concerns about study visit compliance | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only participants receiving study treatment were included in the analysis. For analysis, participants receiving placebo (of any dose-volume equivalent) are pooled within arm per the pre-specified analysis plan.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm A: 0 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236 | Arm C: 0 mg/kg SAR441236 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 10 | 10 | 5 | 2 | 4 | 4 | 4 | 51
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [51 to 55] | 47 [32 to 57] | 51 [41 to 56] | 51 [37 to 57] | 57 [54 to 60] | 26 [25 to 30] | 25 [24 to 26] | 54 [50 to 63] | 54 [39 to 62] | 53 [49 to 57] | 53 [37 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5
  Male | 4 | 2 | 3 | 9 | 10 | 5 | 2 | 4 | 3 | 4 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White (Non-Hispanic) | 3 | 2 | 2 | 3 | 6 | 3 | 0 | 3 | 1 | 1 | 24
  Race/Ethnicity: Black (Non-Hispanic) | 1 | 2 | 2 | 6 | 1 | 1 | 2 | 1 | 2 | 1 | 19
  Race/Ethnicity: Hispanic or Latino (regardless of race) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 6
  Race/Ethnicity: Other (Non-Hispanic) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
HIV RNA [Count of Participants; unit: Participants] — Population: HIV RNA categories for ART-suppressed participants in Arms A and C only.
  Participants
    number analyzed (Participants) | 4 | 4 | 4 | 10 | 10 | 0 | 0 | 4 | 4 | 4 | 44
    <40 copies/mL | 4 | 4 | 4 | 8 | 10 |  |  | 4 | 4 | 4 | 42
    ≥40 copies/mL | 0 | 0 | 0 | 2 | 0 |  |  | 0 | 0 | 0 | 2
HIV RNA [Count of Participants; unit: Participants] — Population: HIV RNA categories for viremic participants in Arm B only.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 0 | 7
    10,000-29,000 copies/mL |  |  |  |  |  | 1 | 0 |  |  |  | 1
    30,000-99,999 copies/mL |  |  |  |  |  | 3 | 1 |  |  |  | 4
    100,000-200,000 copies/mL |  |  |  |  |  | 0 | 1 |  |  |  | 1
    ≥200,000 copies/mL |  |  |  |  |  | 1 | 0 |  |  |  | 1
CD4 Cell Count [Count of Participants; unit: Participants]
  250-499 cells/mm^3 | 0 | 2 | 0 | 3 | 3 | 2 | 2 | 1 | 0 | 1 | 14
  ≥500 cells/mm^3 | 4 | 2 | 4 | 7 | 7 | 3 | 0 | 3 | 4 | 3 | 37
Baseline Weight [Median (Inter-Quartile Range); unit: kilograms] | 91 [88 to 98] | 83 [80 to 97] | 96 [76 to 102] | 83 [75 to 89] | 88 [86 to 95] | 67 [66 to 78] | 83 [69 to 98] | 86 [79 to 91] | 97 [93 to 104] | 82 [72 to 88] | 87 [77 to 94]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Experiencing a Grade 3 or Higher Adverse Event (AE) That is Related to Study Treatment.
Description: The proportion of participants reporting a grade 3 (severe), grade 4 (potentially life-threatening), or grade 5 (death) adverse event, that was judged by the core safety team (blinded to active/placebo treatment in Arms A and C) to be at least possibly related to study treatment.
  Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017
Time Frame: Measured from Day 0 through entire study follow-up, up to 24 weeks post study treatment administration for single dose cohorts (all arms) and up to 36 weeks after the fourth study treatment administration for the multi-dose cohort (Arm A only).
Population: All participants exposed to SAR441236/placebo. Those receiving placebo of any dose-volume equivalent are pooled w/in arm per the analysis plan. The highest dose in ArmA (Cohort 4) was designed to with dual safety objectives: 1) evaluate the safety of a single dose for 12 weeks and 2) evaluate the safety of multiple doses if the initial dose proved safe.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm A: 0 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236 | Arm C: 0 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 10 | 10 | 5 | 2 | 4 | 4 | 4
Proportion of participants | 0 [0 to 0.60] | 0 [0 to 0.60] | 0 [0 to 0.60] | 0 [0 to 0.31] | 0 [0 to 0.31] | 0 [0 to 0.52] | 0 [0 to 0.84] | 0 [0 to 0.6] | 0 [0 to 0.6] | 0 [0 to 0.6]

2. Primary Outcome: Mean Dose-normalized AUC 0-12wk of SAR441236
Description: Dose-normalized Area Under the Concentration time curve (AUC) for each participant was calculated from all available SAR441236 concentrations measured prior to and after first treatment and prior to any subsequent treatment instances (Arm A: 30 mg/kg only). Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine AUC 0-12WK.
Time Frame: SAR441236 PK samples at pre-dose, Hours 0, 2 (Arm A, B only) , 4 (Arm A, B only), 6 (Arm A, B only), and 10, Days 1, 2, 3, 4 (Arm B only), 7, 10 (Arm B only), and Weeks 2, 4, 8 (single dose only), 10 (multi dose only), and 12.
Population: All participants who have been exposed to SAR441236 and have evaluable levels of SAR441236 such that AUC 0-12WK can be calculated.
Measure: Median (Standard Error); unit: (ug*day/mL)/(mg/kg)
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 7 | 1 | 1 | 4 | 4
(ug*day/mL)/(mg/kg) | 593 (282) | 631 (120) | 610 (54.5) | 743 (296) | 552 | 159 | 254 (145) | 236 (126)
Statistical Analysis 1: Comparison: Arm A: 1 mg/kg SAR441236 vs Arm A: 3 mg/kg for SAR441236 vs Arm A: 10 mg/kg SAR441236 vs Arm A: 30 mg/kg SAR441236 vs Arm C: 0.3 mg/kg SAR441236 vs Arm C: 1 mg/kg SAR441236; As dose-normalized AUC 0-12WK values were considered, participants were pooled within Arm (i.e., Arm A participants receiving 1, 3, 10, or 30 mg/kg were pooled and Arm C participants 0.3 or 1.0 mg/kg were pooled); Test type: Equivalence — Confidence Interval (CI) on Geometric Mean Ratio; Geometric Mean Ratio = 3.2, 95% CI 2-sided [1.9 to 5.3] — The ratios of the geometric means (Arm A/Arm C) and the corresponding 95% CI were obtained by exponentiating the least squares mean difference and its 95% CI of the natural log-transformed data; No comparisons were done with Arm B participants, as only two participants in that arm had available measurements such that AUC 0-12WK could be estimated

3. Primary Outcome: Mean Change in Plasma HIV-1 RNA (log10 Copies/mL) From Baseline to Day 7 of SAR441236 Monotherapy for Viremic Participants With HIV (Arm B Cohorts)
Description: Baseline was defined as the last measurement taken prior to treatment initiation. Change was calculated as the log10-transformed value on Day 7 minus the log10-transformed value at baseline.
Time Frame: Measured at Day 0 and Day 7
Population: Arm B participants who actually received ≥0.9 mg/kg SAR441236, had an entry plasma HIV-1 RNA ≥ 5000 copies/mL, and had Plasma HIV-1 RNA measured at the scheduled study visits were included.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236
Number analyzed (Participants) | 5 | 2
log10 copies/mL | -0.10 (0.42) | -0.38 (0.24)
Statistical Analysis 1: Comparison: Arm B: 1 mg/kg SAR441236 vs Arm B: 30 mg/kg SAR441236; Arm B participants were pooled across doses for analysis; Test type: Other; p = 0.26, t-test, 2 sided — Under the null hypothesis, it was assumed there was no change in HIV-1 RNA (log10 copies/mL) from baseline to Day 7 of SAR441236 monotherapy for viremic participants with HIV (Arm B cohorts); Mean = -0.18, 95% CI 2-sided [-0.53 to 0.18]

4. Secondary Outcome: Mean Change in Plasma HIV-1 RNA (log10 Copies/mL) From Baseline to Post-infusion Time Points During SAR441236 Monotherapy for Viremic Participants With HIV (Arm B Cohorts)
Description: Baseline was defined as the last measurement taken prior to treatment initiation. Change was calculated as the log10-transformed value of plasma HIV-1 RNA at the post-infusion time point minus the log10-transformed value at baseline.
Time Frame: Measured at Day 0 and at Day 1, 2, 3, and 4, and Week 1, 2, and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236
Number analyzed (Participants) | 5 | 2
log10 copies/mL
  Change from baseline to Day 1 | 0.04 (0.07) | 0.10 (0.12)
  Change from baseline to Day 2 | 0.04 (0.14) | -0.06 (0.07)
  Change from baseline to Day 3 | -0.04 (0.20) | -0.39 (0.04)
  Change from baseline to Day 4: number analyzed (Participants) | 4 | 2
  Change from baseline to Day 4 | 0.01 (0.40) | -0.68 (0.03)
  Change from baseline to Week 1 | -0.10 (0.42) | -0.38 (0.24)
  Change from baseline to Week 2: number analyzed (Participants) | 4 | 2
  Change from baseline to Week 2 | -0.08 (0.08) | 0.09 (0.38)
  Change from baseline to Week 3: number analyzed (Participants) | 4 | 2
  Change from baseline to Week 3 | 0.03 (0.37) | 0.07 (0.48)

5. Secondary Outcome: Mean Change in Plasma HIV-1 RNA (log10 Copies/mL) From Baseline to Day 14 of SAR441236 Monotherapy for Viremic Participants With HIV (Arm B Cohorts)
Description: Baseline was defined as the last measurement taken prior to treatment initiation. Change was calculated as the value of plasma HIV-1 RNA on Day 14 minus the value at baseline.
Time Frame: Measured at Day 0 and Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Arm B: 30 mg/kg SAR441236: Participants received 1 mg/kg of SAR441236, administered as a single IV infusion on Day 0. Antiretroviral treatment was initiated or re-initiated by Day 28 (Cohort 5).
  SAR441236: Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
Arm/Group | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236
Number analyzed (Participants) | 4 | 2
log10 copies/mL | -0.08 (0.08) | 0.09 (0.38)
Statistical Analysis 1: Comparison: Arm B: 1 mg/kg SAR441236 vs Arm B: 30 mg/kg SAR441236; Arm B participants were pooled across doses for analysis; Test type: Other; p = 0.78, t-test, 2 sided — Under the null hypothesis, it was assumed there was no change in HIV-1 RNA (log10 copies/mL) from baseline to Day 14 of SAR441236 monotherapy for viremic participants with HIV (Arm B cohorts); Mean = -0.02, 95% CI 2-sided [-0.24 to 0.19]

6. Secondary Outcome: Mean Maximum Reduction of Plasma HIV-1 RNA During up to 28 Days of SAR441236 Monotherapy for Viremic Participants With HIV (Arm B Cohorts)
Description: The maximum reduction in plasma HIV-1 RNA was calculated as the largest decline from baseline, defined as the last measurement taken prior to treatment initiation, to any post-infusion timepoint while the participant was on SAR441236 monotherapy (i.e., prior to initiating or reinitiating ART).
Time Frame: Measured at Day 0 and at up to Day 28 (while on SAR441236 monotherapy)
Population: Arm B participants who actually received ≥0.9 mg/kg SAR441236 and had an entry plasma HIV-1 RNA ≥ 5000 copies/mL.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236
Number analyzed (Participants) | 5 | 2
log10 copies/mL | -0.30 (0.23) | -0.68 (0.03)

7. Secondary Outcome: Attributions of Anti-SAR441236 Antibodies Among Participants in Single-dose Cohorts.
Description: Number of participants who were anti-drug antibody (ADA) negative, ADA positive (treatment induced), and missing were calculated at each sampled timepoint.
Time Frame: Measured at Day 0 and at Week 2, 4, 12, and 24
Population: Participants who received SAR441236 (not placebo) were tested for the presence of anti-drug antibodies. Only participants enrolled in single-dose cohorts were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 2 | 4 | 4
Participants
  ADA Status at Day 0: Positive: Treatment-Induced | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Status at Day 0: Negative | 4 | 4 | 4 | 5 | 2 | 4 | 4
  ADA Status at Day 0: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Status at Week 2: Positive: Treatment-Induced | 0 | 0 | 1 | 1 | 1 | 0 | 1
  ADA Status at Week 2: Negative | 4 | 4 | 3 | 3 | 1 | 4 | 3
  ADA Status at Week 2: Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ADA Status at Week 4: Positive: Treatment-Induced | 0 | 0 | 1 | 4 | 0 | 0 | 0
  ADA Status at Week 4: Negative | 3 | 4 | 3 | 1 | 2 | 4 | 4
  ADA Status at Week 4: Missing | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Status at Week 12: Positive: Treatment-Induced | 0 | 1 | 1 | 2 | 0 | 0 | 1
  ADA Status at Week 12: Negative | 4 | 3 | 3 | 0 | 1 | 4 | 3
  ADA Status at Week 12: Missing | 0 | 0 | 0 | 3 | 1 | 0 | 0
  ADA Status at Week 24: Positive: Treatment-Induced | 0 | 1 | 0 | 3 | 0 | 0 | 2
  ADA Status at Week 24: Negative | 4 | 3 | 4 | 0 | 0 | 4 | 2
  ADA Status at Week 24: Missing | 0 | 0 | 0 | 2 | 2 | 0 | 0

8. Secondary Outcome: Attributions of Anti-SAR441236 Antibodies Among Participants in Multi-dose Cohort.
Description: as for outcome 7
Time Frame: Measured at Day 0, at Weeks 2 and 4 after Infusion 1, at Infusion 2, at Infusion 3, at Infusion 4, and at Weeks 12 and 36 post-Infusion 4
Population: Participants who received SAR441236 (not placebo) were tested for the presence of anti-drug antibodies. Only participants enrolled in the multi-dose cohort were included. Samples for one 30 mg/kg SAR441236 were lost in a freezer malfunction and no results were able to be obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 30 mg/kg SAR441236
Number analyzed (Participants) | 9
Participants
  ADA Status at Inf 1: Day 0: Positive: Treatment-Induced | 0
  ADA Status at Inf 1: Day 0: Negative | 9
  ADA Status at Inf 1: Day 0: Missing | 0
  ADA Status at Inf 1: Week 2: Positive: Treatment-Induced | 0
  ADA Status at Inf 1: Week 2: Negative | 8
  ADA Status at Inf 1: Week 2: Missing | 1
  ADA Status at Inf 1: Week 4: Positive: Treatment-Induced | 0
  ADA Status at Inf 1: Week 4: Negative | 7
  ADA Status at Inf 1: Week 4: Missing | 2
  ADA Status at Inf 2: Day 0: Positive: Treatment-Induced | 1
  ADA Status at Inf 2: Day 0: Negative | 5
  ADA Status at Inf 2: Day 0: Missing | 3
  ADA Status at Inf 3: Day 0: Positive: Treatment-Induced | 0
  ADA Status at Inf 3: Day 0: Negative | 6
  ADA Status at Inf 3: Day 0: Missing | 3
  ADA Status at Inf 4: Day 0: Positive: Treatment-Induced | 0
  ADA Status at Inf 4: Day 0: Negative | 6
  ADA Status at Inf 4: Day 0: Missing | 3
  ADA Status at Inf 4: Week 12: Positive: Treatment-Induced | 0
  ADA Status at Inf 4: Week 12: Negative | 6
  ADA Status at Inf 4: Week 12: Missing | 3
  ADA Status at Inf 4: Week 36: Positive: Treatment-Induced | 1
  ADA Status at Inf 4: Week 36: Negative | 4
  ADA Status at Inf 4: Week 36: Missing | 4

9. Secondary Outcome: Mean Change From Baseline in CD4+ T Cell Counts Following the First Treatment of SAR441236 or Placebo for All Cohorts
Description: Baseline was defined as the last measurement obtained prior to treatment initiation. Change was calculated as the value of CD4+ T cell counts (cells/mm^3) at Week 12 (prior to subsequent study treatment, if any) minus the value at baseline.
Time Frame: Measured at Day 0 and Week 12
Population: All participants who received study treatment (SAR441236 or placebo) and had CD4 counts measured at the scheduled study visits were included.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm A: 0 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236 | Arm C: 0 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 3 | 9 | 10 | 2 | 1 | 4 | 4 | 4
cells/mm^3 | -6 (87) | -96 (222) | 96 (249) | -36 (246) | -43 (117) | 10 (273) | 138 (NA) — No standard deviation due to N=1 | 61 (176) | -136 (216) | -53 (289)

10. Secondary Outcome: Mean Change From Baseline in CD4+ T Cell Counts Following Each Infusion for Cohort 4
Description: Baseline was defined as the last measurement obtained prior to treatment initiation. Change was calculated as the value of CD4 + T cell counts (cells/mm^3) at Week 12 after each infusion minus the value at baseline.
Time Frame: Measured at Day 0 and at Week 12 after each infusion
Population: Arm A participants who received multiple infusions (SAR441236 or placebo) and had CD4 count measured at the scheduled study visits were included.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- Arm A: 0 mg/kg SAR441236: Placebo participants were pooled across those receiving:
  • 30 mg/kg dose volume-equivalent administered as an IV infusion on Day 0 and then every 12 weeks for a total of four doses (Cohort 4)
  All continued on non-study provided ART.
  Placebo: Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
Arm/Group | Arm A: 30 mg/kg SAR441236 | Arm A: 0 mg/kg SAR441236
Number analyzed (Participants) | 6 | 4
cells/mm^3
  Change in from baseline to Week 12 after 2nd treatment | 73 (357) | 28 (190)
  Change in from baseline to Week 12 after 3rd treatment | 78 (232) | 17 (252)
  Change in from baseline to Week 12 after 4th treatment | -83 (253) | 77 (111)

11. Secondary Outcome: Mean Maximum Concentration (Cmax) of SAR441236 After a Single IV Infusion or SC Injection.
Description: Cmax for each participant was calculated as the maximum observed concentration from all available SAR441236 concentrations measured prior to and after first treatment and prior to any subsequent treatment instances (Arm A: 30 mg/kg only). Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine Cmax.
Time Frame: SAR441236 PK samples at pre-dose, Hours 0, 2 (Arm A, B only) , 4 (Arm A, B only), 6 (Arm A, B only), and 10, Days 1, 2, 3, 4 (Arm B only), 7, 10 (Arm B only), and Weeks 2, 4, 8 (single dose only), 10 (multi dose only), 12, and 24 (single dose only).
Population: All participants exposed to SAR441236 with evaluable levels of SAR441236 such that Cmax can be derived.
Measure: Mean (Standard Error); unit: (ug/mL)
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 9 | 5 | 2 | 4 | 4
(ug/mL) | 25.2 (11) | 72.7 (27.7) | 295 (265) | 771 (250) | 24.9 (3.5) | 483 (249) | 1.69 (0.74) | 4.77 (2.32)

12. Secondary Outcome: Half-life (T1/2) of SAR441236 After a Single IV Infusion or SC Injection.
Description: Half-life for each participant was calculated using regression analysis on all available SAR441236 concentrations measured prior to and after first treatment and prior to any subsequent treatment instances (Arm A: 30 mg/kg only). Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine half-life.
Time Frame: as for outcome 11
Population: All participants exposed to SAR441236 with evaluable levels of SAR441236 such that half-life can be derived.
Measure: Mean (Standard Deviation); unit: (days)
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 9 | 5 | 2 | 4 | 4
(days) | 34.8 (4.73) | 38.1 (4.94) | 30.9 (4.90) | 37.0 (6.46) | 27.2 (2.37) | 23.2 (3.97) | 58.5 (1.41) | 47.7 (6.13)

13. Secondary Outcome: Time to Maximum Concentration (Tmax) of SAR441236 After a Single IV Infusion of SC Injection.
Description: Tmax for each participant was time to maximum observed SAR441236 measured from all available SAR441236 concentrations measured prior to and after first treatment and prior to any subsequent treatment instances (Arm A: 30 mg/kg only). Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine Tmax.
Time Frame: as for outcome 11
Population: All participants exposed to SAR441236 with evaluable levels of SAR441236 such that Cmax, and corresponding Tmax, can be derived.
Measure: Mean (Standard Error); unit: (days)
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 9 | 5 | 2 | 4 | 4
(days) | 0.07 (0.05) | 2.11 (4.06) | 0.12 (0.08) | 0.16 (0.15) | 0.09 (0.12) | 0.09 (0.06) | 6.71 (5.19) | 5.07 (2.49)

14. Secondary Outcome: Clearance or Apparent Clearance of SAR441236 After a Single IV Infusion of SC Injection.
Description: Clearance (CL, in Arms A and B) or Apparent Clearance (CL/F, in Arm C) for each participant was calculated from all available SAR441236 concentrations measured prior to and after first treatment and prior to any subsequent treatment instances (Arm A: 30 mg/kg only). Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine CL and CL/F.
Time Frame: as for outcome 11
Population: All participants exposed to SAR441236 with evaluable levels of SAR441236 such that clearance (Arms A and B) or apparent clearance (Arm C) can be derived.
Measure: Mean (Standard Deviation); unit: (mL/day)
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 9 | 5 | 2 | 4 | 4
(mL/day) | 181 (148) | 116 (14.9) | 130 (43.5) | 122 (50.2) | 132 (28.1) | 348 (51.6) | 163 (36.0) | 399 (318)

15. Secondary Outcome: Volume of Distribution of SAR441236 After a Single IV Infusion or SC Injection
Description: Volume of distribution (Arms A and B) or apparent volume of distribution (Arm C) was calculated from all available SAR441236 concentrations measured prior to and after first treatment and prior to any subsequent treatment instances (Arm A: 30 mg/kg only). Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine volume of distribution and apparent volume of distribution.
Time Frame: as for outcome 11
Population: All participants exposed to SAR441236 with evaluable levels of SAR441236 such that volume of distribution (Arms A and B) or apparent volume of distribution (Arm C) can be derived.
Measure: Mean (Standard Deviation); unit: (L)
Arm/Group | Arm A: 1 mg/kg SAR441236 | Arm A: 3 mg/kg for SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236
Number analyzed (Participants) | 4 | 4 | 4 | 9 | 5 | 2 | 4 | 4
(L) | 8.02 (3.13) | 5.90 (1.56) | 5.34 (0.48) | 5.96 (1.05) | 5.27 (0.79) | 9.73 (0.38) | 14.0 (2.79) | 22.8 (14.7)

16. Secondary Outcome: Mean Maximum Concentration (Cmax) of SAR441236 After the Fourth IV Infusion
Description: Cmax after the fourth infusion was calculated as the maximum observed SAR441236 concentration from SAR441236 PK samples obtained after the fourth infusion. Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine Cmax after the 4th infusion.
Time Frame: Intensive SAR441236 PK samples after Infusion 4 (Week 36) at Hours 0, 2, 4, 6, and 10, Days 1 and 2, and at non-intensive sampling at Weeks 37, 38, 40, 48, 60, and 72.
Population: All participants exposed to 4 infusions of SASR441236 (30 mg/kg participants only) with evaluable levels of SAR441236 such that Cmax can be derived.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm A: 30 mg/kg SAR441236
Number analyzed (Participants) | 6
ug/mL | 890.50 (176.66)

17. Secondary Outcome: Mean SAR441236 Concentration 12 Weeks After Infusions 1, 2, 3, and 4
Description: SAR441236 concentration for each participant was calculated as the observed SAR441236 concentration 12 weeks after each infusion.
Time Frame: SAR441236 PK samples at Week 12, 24, 36, and 48.
Population: All participants exposed to 4 infusions of SAR441236 (30 mg/kg participants only) with evaluable levels of SAR441236. Only participants who maintained the every 12-week dosing schedule were considered for concentration levels 12 weeks after infusions 2-4.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm A: 30 mg/kg SAR441236
Number analyzed (Participants) | 6
ug/mL
  SAR441236 Concentration at Infusion 1 + 12 Weeks | 88.28 (46.73)
  SAR441236 Concentration at Infusion 2 + 12 Weeks: number analyzed (Participants) | 3
  SAR441236 Concentration at Infusion 2 + 12 Weeks | 136.87 (48.78)
  SAR441236 Concentration at Infusion 3 + 12 Weeks: number analyzed (Participants) | 3
  SAR441236 Concentration at Infusion 3 + 12 Weeks | 120.00 (40.84)
  SAR441236 Concentration at Infusion 4 + 12 Weeks: number analyzed (Participants) | 3
  SAR441236 Concentration at Infusion 4 + 12 Weeks | 122.40 (45.43)

18. Secondary Outcome: Mean AUC After Multiple Infusions of SAR441236
Description: Area Under the Concentration time curve (AUC) for multiple infusions of SAR441236 was calculated using all available SAR441236 concentrations. Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine AUC.
Time Frame: Intensive SAR441236 PK samples taken at Hours 0, 2, 4, 6, and 10 and Days 1 and 2 after infusions 1 and 4 and non-intensive sampling at pre-dose (Weeks 0, Week 12, 24, 36) and Weeks 2, 4 , 8, 10, 13, 14, 16, 22, 26, 28, 34, 37, 38, 40, and 48.
Population: All participants exposed to 4 infusions of SAR441236 (30 mg/kg participants only) with evaluable levels of SAR441236. Only participants who maintained the every 12-week dosing schedule were considered for AUC12-24WK, AUC 24-36 WK, AUC 36-48 WK, and AUC 0-48 WK.
Measure: Mean (Standard Deviation); unit: (ug*day)/mL
Arm/Group | Arm A: 30 mg/kg SAR441236
Number analyzed (Participants) | 3
(ug*day)/mL
  AUC 12-24 Week | 26508.02 (5914.53)
  AUC 24-36 Week | 21809.83 (7210.58)
  AUC 36-48 Week | 26137.06 (5336.72)
  AUC 0-48 Week | 96277.43 (17105.70)

19. Secondary Outcome: Mean AUC Accumulation Index (AI) (12 Weeks Post-Dose 1 vs 12 Weeks Post-Dose 4).
Description: The AUC AI (12 Weeks post-Dose 1 vs 12 Weeks post-Dose 4) was calculated as the ratio of AUC 36-48 Weeks and AUC 0-12 Weeks. Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine AUC AI.
Time Frame: as for outcome 18
Population: All participants exposed to 4 infusions of SAR441236 (30 mg/kg participants only) with evaluable levels of SAR441236. Only participants who maintained the every 12-week dosing schedule were considered for AUC AI.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A: 30 mg/kg SAR441236
Number analyzed (Participants) | 3
Ratio | 1.24 (0.18)

20. Secondary Outcome: Mean Trough Accumulative Index (12 Weeks Post-Dose 1 vs 12 Weeks Post-Dose 4)
Description: The Trough AI was calculated as the ratio of the SAR441236 concentration observed 12 weeks after the 4th dose and the SAR441236 concentration observed 12 weeks after the 1st dose. Standard noncompartmental techniques, using Phoenix WinNonlin, were used to determine trough AI.
Time Frame: SAR441236 PK samples taken at Week 12 (pre-dose #2) and at Week 48 (12 weeks after dose #4)
Population: All participants exposed to 4 infusions of SAR441236 (30 mg/kg participants only) with evaluable levels of SAR441236. Only participants who maintained the every 12-week dosing schedule were considered for Trough AI (Dose 1 vs Dose 4)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A: 30 mg/kg SAR441236
Number analyzed (Participants) | 3
Ratio | 1.13 (0.04)

21. Secondary Outcome: Dose-response Relationship Between SAR441236 Exposure and Changes in Plasma HIV-1 RNA
Description: This relationship is based on measured SAR441236 concentrations and HIV-1 RNA values prior to participants initiating ART.
Time Frame: Day 0 and at all study visits prior to ART initiation/re-initiation (up to Week 4)
Population: Only Arm B participants (who were off ART and viremic at entry) were considered for this outcome. Summaries of viral response are provided in outcomes 3, 4, 5, and 6. However, the dose-response relationship cannot be modeled due to insufficient sample size.
Arm/Group | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From study entry to study completion (36 weeks after the final infusion for Cohort 4 and 24 weeks after the first infusion/injection for other cohorts) or premature study discontinuation.
Description: The DAIDS Adverse Event Grading Table(V2.1), July 2017 was used. Participants receiving placebo are pooled w/in arm per the analysis plan. AEs were recorded if:
  * Grade ≥2 AE
  * Any AE leading to change in study treatment
  * AE meeting the Serious Adverse Event definition or Expedited Adverse Event reporting requirement
  * Grade ≥1 rash, urticaria, angioedema, ALT, AST, WBC counts, eosinophilia, AIDS-defining illness, or lab finding the day of or w/in 2 wks of treatment administration
Groups:
- Arm A: 1mg/kg SAR441236: Participants continued on non-study-provided ART and received 1 mg/kg of SAR441236, administered as a single intravenous (IV) infusion on Day 0 (Cohort 1).
  SAR441236: Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
- Arm A: 3 mg/kg SAR441236: Experimental: Arm A: 3 mg/kg SAR441236 Participants continued on non-study-provided ART, and received 3 mg/kg of SAR441236, administered as a single IV infusion on Day 0 (Cohort 2).
  SAR441236: Administered by intravenous (IV) infusion(s) or subcutaneous (SC) injection(s)
Arm/Group | Arm A: 1mg/kg SAR441236 | Arm A: 3 mg/kg SAR441236 | Arm A: 10 mg/kg SAR441236 | Arm A: 30 mg/kg SAR441236 | Arm A: 0 mg/kg SAR441236 | Arm B: 1 mg/kg SAR441236 | Arm B: 30 mg/kg SAR441236 | Arm C: 0.3 mg/kg SAR441236 | Arm C: 1 mg/kg SAR441236 | Arm C: 0 mg/kg SAR441236
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/11 | 0/10 | 0/5 | 0/2 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 0/4 | 2/11 | 0/10 | 1/5 | 0/2 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 4/4 | 3/4 | 8/11 | 8/10 | 5/5 | 0/2 | 1/4 | 3/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 1mg/kg SAR441236 (N=4) | Arm A: 3 mg/kg SAR441236 (N=4) | Arm A: 10 mg/kg SAR441236 (N=4) | Arm A: 30 mg/kg SAR441236 (N=11) | Arm A: 0 mg/kg SAR441236 (N=10) | Arm B: 1 mg/kg SAR441236 (N=5) | Arm B: 30 mg/kg SAR441236 (N=2) | Arm C: 0.3 mg/kg SAR441236 (N=4) | Arm C: 1 mg/kg SAR441236 (N=4) | Arm C: 0 mg/kg SAR441236 (N=4)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 1mg/kg SAR441236 (N=4) | Arm A: 3 mg/kg SAR441236 (N=4) | Arm A: 10 mg/kg SAR441236 (N=4) | Arm A: 30 mg/kg SAR441236 (N=11) | Arm A: 0 mg/kg SAR441236 (N=10) | Arm B: 1 mg/kg SAR441236 (N=5) | Arm B: 30 mg/kg SAR441236 (N=2) | Arm C: 0.3 mg/kg SAR441236 (N=4) | Arm C: 1 mg/kg SAR441236 (N=4) | Arm C: 0 mg/kg SAR441236 (N=4)
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal foot infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 5 | 1 | 2 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 1
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 2 | 2 | 6 | 8 | 4 | 0 | 0 | 2 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The dosing schedule for many Arm A Cohort 4 participants was interrupted by the COVID-19 pandemic and associated study pause. Enrollment in Arm B was limited. Protocol V3.0 closed the 1 mg/kg cohort and opened the 30 mg/kg cohort. Protocol V4.0 modified the eligibility criteria to boost enrollment but, despite the study remaining open through April 2023, no more participants enrolled. Neither Arm B cohort fully enrolled and the intermediate dose cohorts (3 and 10 mg/kg) did not open.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form: Protocol Version 4.0 (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03705169/Prot_ICF_000.pdf
  • Study Protocol: Clarification Memo 1 (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03705169/Prot_001.pdf
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03705169/SAP_002.pdf